CLINICAL TRIAL: NCT01397734
Title: Targeting of the Leukemia Stem Cell Population With Arsenic Trioxide and Tyrosine Kinase Inhibitors for CML
Brief Title: Arsenic Trioxide and Tyrosine Kinase Inhibitors for Chronic Myelogenous Leukemia (CML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment and limited funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, David Avigan, MD, Prinicipal Investigator, Beth Israel Deaconess Medical Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-107
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: CML; Chronic myelogenous leukemia; Chronic Myeloid leukemia; Arsenic; Arsenic trioxide; Imatinib; Dasatinib; Nilotinib; TKI; Tyrosine kinase inhibitor
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Patients who are receiving Imatinib as part of their standard of care therapy for CML.
  Interventions: Drug: Arsenic trioxide
- Cohort 2 (Experimental): Patients who are receiving Dasatinib as part of their standard of care therapy for CML.
  Interventions: Drug: Arsenic trioxide
- Cohort 3 (Experimental): Patients who are receiving Nilotinib as part of their standard of care therapy for CML.
  Interventions: Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Arsenic trioxide — 0.15mg/kg/day Arsenic trioxide given IV on days 1-5 of the cycle.

SUMMARY:
In this research study, the investigators are looking to see whether the combination of arsenic trioxide with a tyrosine kinase inhibitor is safe, and what effects it has on chronic myelogenous leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of chronic myelogenous leukemia as confirmed by fluorescent In Situ Hybridization (FISH) for BCR/ABL translocation and/or standard cytogenetics analysis.
* Participants may have received prior hydroxyurea but may not be currently being treated with hydroxyurea at the time of study initiation.
* Participants may have received prior TKI therapy, however must be on a stable dose of their current TKI for at least one month prior to enrollment.
* Participants must demonstrate evidence of persistent disease either by cytogenetics/FISH or by PCR for BCR/ABL in the peripheral blood or bone marrow.
* Greater than or equal to 18 years in age. Because little dosing or adverse event data are currently available on the use of Arsenic in participants <18 years of age, children are excluded from this study.
* Life expectancy of greater than 3 months
* ECOG performance status <2
* Participants must have normal organ and marrow function as defined below:

  * Bilirubin ≤ 2.0 mg/dL
  * Creatinine ≤ 2 mg/dL
  * ALT < 2.5 X institutional upper limit of normal
  * AST < 2.5 X institutional upper limit of normal
  * WBC > 2.0 K/uL
  * Platelets >100K
* Oxygen saturation > 95% on room air
* The effects of Arsenic on the developing human fetus are unknown. For this reason, women of child-bearing potential must have a documented negative pregnancy test; in addition, agreement to use adequate contraception (hormonal or barrier method of birth control; abstinence) must be documented for both women of child-bearing potential and men prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* All patients must demonstrate the ability to understand the investigational nature of this study and must sign a written informed consent document in accordance with institutional and federal guidelines

Exclusion Criteria:

* History of acute myocardial infarction, unstable angina, congestive heart failure, or arrhythmia within the last three months
* Participants may not be receiving any other study agent
* Mean QTc> 450 ms at time of screening
* Use of potassium wasting diuretics during study treatment
* Patients should not be taking drugs that are generally accepted to have a risk of causing Torsades de Pointes. The following must be discontinued at least 7 days prior to enrollment to be eligible: quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Drugs that are highly dependent on CYP3A4 for metabolism and have a narrow therapeutic index (see Appendix A) are allowed but must be used with caution
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Concurrent and or uncontrolled psychiatric or medical condition which may interfere with the study completion.
* Pregnant women are excluded from this study because the risk of Arsenic to a developing fetus is unknown. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with Arsenic, breastfeeding should be discontinued if the mother is treated on this clinical trial
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with TKI therapy and Arsenic. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-09; Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Toxicity | 1, 2, 6, 12 months
  To assess the safety and toxicity of arsenic in combination with TKI therapy for chronic phase CML patients

SECONDARY OUTCOMES:
Disease Response | 1, 2, 6, 12 months
  To assess disease response after combined therapy arsenic trioxide and imatinib (cohort 1), dasatinib (cohort 2) or nilotinib (cohort 3) by bone marrow cytogenetic assessment and serial BCR-ABL QPCR from peripheral blood and bone marrow measurements. Rates of major and complete cytogenetic and molecular responses will be determined.
PML Expression | 1, 6, 12 months
  To assess whether combined therapy with arsenic and imatinib, dasatinib or nilotinib results in decreased PML expression on the CML stem cell compartment, and decreased capacity of CML stem cells to maintain long term proliferative capacity.

CONTACTS AND LOCATIONS:
Overall Officials: David E Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States